CLINICAL TRIAL: NCT03038620
Title: Impact of Liraglutide 3.0 on Body Fat Distribution, Visceral Adiposity, and Cardiometabolic Risk Markers In Overweight and Obese Adults at High Risk for Cardiovascular Disease
Brief Title: Impact of Liraglutide 3.0 on Body Fat Distribution
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Parag Joshi, M.D., University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU 122015-044
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Obesity, Visceral; Cardiovascular Diseases; Fat Disorder
Keywords: Obesity; Visceral; Cardiovascular Disease; Fat
MeSH Terms: conditions — Obesity, Abdominal; Cardiovascular Diseases; Lipid Metabolism Disorders; Obesity; Platelet Glycoprotein IV Deficiency | interventions — Liraglutide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liraglutide 3.0 mg (Experimental): Drug: Liraglutide Active Drug
  Other Names:
  * Saxenda
  Escalate the liraglutide (active) dose to 3.0 mg/day over a 4 week period following an initial dose of 0.6 mg/day and weekly dose escalation steps of 0.6 mg/day through subcutaneous injection.
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Drug: Placebo (for Liraglutide at a concentration of 6.0 mg/mL) Placebo tablet manufactured to mimic Liraglutide at a concentration of 6.0 mg/mL
  Other Names:
  * Placebo
  * Saline injection
  Escalate the Placebo dose to 3.0 mg/day over a 4 week period following an initial dose of 0.6 mg/day and weekly dose escalation steps of 0.6 mg/day through subcutaneous injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Liraglutide is administered once daily by subcutaneous injections with the pen-injector, either in the abdomen, thigh or upper arm. Injections can be done at any time of day irrespective of meals. Subjects will be instructed to escalate the liraglutide dose to 3.0 mg/day over a 4 week period following an initial dose of 0.6 mg/day and weekly dose escalation steps of 0.6 mg/day.
  Other Names: Saxenda
  Arms: Liraglutide 3.0 mg
Drug: Placebo — Placebo is administered once daily by subcutaneous injections with the pen-injector, either in the abdomen, thigh or upper arm. Injections can be done at any time of day irrespective of meals. Subjects will be instructed to escalate the placebo dose to 3.0 mg/day over a 4 week period following an initial dose of 0.6 mg/day and weekly dose escalation steps of 0.6 mg/day.
  Other Names: Saline injection
  Arms: Placebo

SUMMARY:
This study is a clinical study to investigate the efficacy of liraglutide compared to placebo in reducing visceral adiposity measured by MRI in overweight or obese subjects at high risk for cardiovascular disease after 40 weeks on-treatment.

DETAILED DESCRIPTION:
Obesity has long been recognized as a risk factor for all-cause mortality and morbidity, including the development of cardiovascular and metabolic diseases such as coronary artery disease, hypertension, insulin resistance, diabetes, and dyslipidemia. Obesity has recently been formally defined as a chronic disease characterized by pathophysiological processes that result in increased adipose tissue mass and can result in increased morbidity and mortality. Although the health risks associated with obesity are clear, there is an emerging appreciation that obesity per se, as defined by simple anthropometric measures such as waist circumference or body mass index (BMI), is neither necessary nor sufficient to promote cardiometabolic disease and atherosclerotic cardiovascular disease (ASCVD) risk. As a result, BMI alone is an insufficient marker of risk and may not accurately identify individuals at elevated risk for ASCVD. There is a pressing need to more accurately phenotype obesity to identify individuals at elevated risk for ASCVD that may benefit from more intensive preventive and therapeutic strategies

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 35 years
* Able to provide informed consent
* BMI ≥ 30 kg/m2 or ≥ 27 kg/m2 with metabolic syndrome
* Metabolic syndrome is defined as at least three of the following:3

  1. waist circumference > 102 cm (40 in) in men and 88 cm (35 in) in women
  2. triglycerides > 150 mg/dL or on treatment for hypertriglyceridemia
  3. HDL cholesterol < 40 mg/dL in men and < 50 mg/dL in women
  4. blood pressure > 130/85 mmHg or on treatment for hypertension
  5. fasting glucose > 100 mg/dL

Exclusion Criteria:

* Treatment with Glucagon-like peptide-1 (GLP-1) receptor agonists (including liraglutide, exenatide or others as they become available), dipeptidyl peptidase 4 (DPP-4) inhibitors or insulin within the last 3 months.
* Receipt of any anti-obesity drug or supplement within 1 month prior to screening for this trial.
* Self-reported or clinically documented history of significant fluctuations (>5% change) in weight within 3 months prior to screening for this trial.
* History of diabetes mellitus (type 1 or 2) or on treatment with anti-diabetes medication.
* History of chronic pancreatitis or idiopathic acute pancreatitis (current or prior history).
* History of gallbladder disease (cholelithiasis or cholecystitis).
* Chronic kidney disease stage III or greater (eGFR<60 mL/min).
* Obesity induced by other endocrinologic disorders (e.g. Cushing Syndrome).
* Current or history of treatment with medications that may cause significant weight gain, within 1 month prior to screening for this trial, including systemic corticosteroids (except for a short course of treatment, i.e., 7- 10 days), tri-cyclic antidepressants, atypical antipsychotic and mood stabilizers (e.g., imipramine, amitryptiline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproic acid and its derivatives, and lithium).
* Diet attempts using herbal supplements or over-the-counter medications within 1 month prior to screening for this trial.
* Current participation in an organized weight reduction program or within the last 1 month prior to screening for this trial.
* Participation in a clinical trial within the last 3 months prior to screening for this trial.
* Familial or personal history of multiple endocrine neoplasia type 2 or familial medullary thyroid carcinoma.
* Personal history of non-familial medullary thyroid carcinoma.
* History of Major Depressive Disorder within the last 2 years.
* History of other severe psychiatric disorders, e.g., schizophrenia, bipolar disorder.
* Any lifetime history of a suicide attempt.
* A history of any suicidal behavior in the last month prior to randomization.
* Surgery scheduled for the trial duration period, except for minor surgical procedures, at the discretion of the Investigator.
* Known or suspected hypersensitivity to trial product(s) or related product(s).
* Known or suspected abuse of alcohol or narcotics.
* Language barrier, mental incapacity, unwillingness or inability to understand.
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods. These include abstinence and the following methods: diaphragm with spermicide, condom with spermicide (by male partner), intrauterine device, sponge, spermicide, Norplant®, Depo-Provera® or oral contraceptives.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parag Joshi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Astrup A, Rossner S, Van Gaal L, Rissanen A, Niskanen L, Al Hakim M, Madsen J, Rasmussen MF, Lean ME; NN8022-1807 Study Group. Effects of liraglutide in the treatment of obesity: a randomised, double-blind, placebo-controlled study. Lancet. 2009 Nov 7;374(9701):1606-16. doi: 10.1016/S0140-6736(09)61375-1. Epub 2009 Oct 23. PMID 19853906
- [Background] Astrup A, Carraro R, Finer N, Harper A, Kunesova M, Lean ME, Niskanen L, Rasmussen MF, Rissanen A, Rossner S, Savolainen MJ, Van Gaal L; NN8022-1807 Investigators. Safety, tolerability and sustained weight loss over 2 years with the once-daily human GLP-1 analog, liraglutide. Int J Obes (Lond). 2012 Jun;36(6):843-54. doi: 10.1038/ijo.2011.158. Epub 2011 Aug 16. PMID 21844879
- [Background] Grundy SM, Cleeman JI, Daniels SR, Donato KA, Eckel RH, Franklin BA, Gordon DJ, Krauss RM, Savage PJ, Smith SC Jr, Spertus JA, Fernando Costa. Diagnosis and management of the metabolic syndrome: an American Heart Association/National Heart, Lung, and Blood Institute scientific statement: Executive Summary. Crit Pathw Cardiol. 2005 Dec;4(4):198-203. doi: 10.1097/00132577-200512000-00018. No abstract available. PMID 18340209
- [Background] Berrington de Gonzalez A, Hartge P, Cerhan JR, Flint AJ, Hannan L, MacInnis RJ, Moore SC, Tobias GS, Anton-Culver H, Freeman LB, Beeson WL, Clipp SL, English DR, Folsom AR, Freedman DM, Giles G, Hakansson N, Henderson KD, Hoffman-Bolton J, Hoppin JA, Koenig KL, Lee IM, Linet MS, Park Y, Pocobelli G, Schatzkin A, Sesso HD, Weiderpass E, Willcox BJ, Wolk A, Zeleniuch-Jacquotte A, Willett WC, Thun MJ. Body-mass index and mortality among 1.46 million white adults. N Engl J Med. 2010 Dec 2;363(23):2211-9. doi: 10.1056/NEJMoa1000367. PMID 21121834
- [Background] Despres JP. Body fat distribution and risk of cardiovascular disease: an update. Circulation. 2012 Sep 4;126(10):1301-13. doi: 10.1161/CIRCULATIONAHA.111.067264. No abstract available. PMID 22949540
- [Background] Garvey WT, Garber AJ, Mechanick JI, Bray GA, Dagogo-Jack S, Einhorn D, Grunberger G, Handelsman Y, Hennekens CH, Hurley DL, McGill J, Palumbo P, Umpierrez G; The Aace Obesity Scientific Committee. American association of clinical endocrinologists and american college of endocrinology position statement on the 2014 advanced framework for a new diagnosis of obesity as a chronic disease. Endocr Pract. 2014 Sep;20(9):977-89. doi: 10.4158/EP14280.PS. No abstract available. PMID 25253227
- [Background] Morkedal B, Vatten LJ, Romundstad PR, Laugsand LE, Janszky I. Risk of myocardial infarction and heart failure among metabolically healthy but obese individuals: HUNT (Nord-Trondelag Health Study), Norway. J Am Coll Cardiol. 2014 Mar 25;63(11):1071-8. doi: 10.1016/j.jacc.2013.11.035. Epub 2013 Dec 15. PMID 24345592
- [Background] Despres JP, Lemieux I, Bergeron J, Pibarot P, Mathieu P, Larose E, Rodes-Cabau J, Bertrand OF, Poirier P. Abdominal obesity and the metabolic syndrome: contribution to global cardiometabolic risk. Arterioscler Thromb Vasc Biol. 2008 Jun;28(6):1039-49. doi: 10.1161/ATVBAHA.107.159228. Epub 2008 Mar 20. PMID 18356555
- [Background] McLaughlin T, Lamendola C, Liu A, Abbasi F. Preferential fat deposition in subcutaneous versus visceral depots is associated with insulin sensitivity. J Clin Endocrinol Metab. 2011 Nov;96(11):E1756-60. doi: 10.1210/jc.2011-0615. Epub 2011 Aug 24. PMID 21865361
- [Background] McLaughlin T, Sherman A, Tsao P, Gonzalez O, Yee G, Lamendola C, Reaven GM, Cushman SW. Enhanced proportion of small adipose cells in insulin-resistant vs insulin-sensitive obese individuals implicates impaired adipogenesis. Diabetologia. 2007 Aug;50(8):1707-15. doi: 10.1007/s00125-007-0708-y. Epub 2007 Jun 5. PMID 17549449
- [Background] See R, Abdullah SM, McGuire DK, Khera A, Patel MJ, Lindsey JB, Grundy SM, de Lemos JA. The association of differing measures of overweight and obesity with prevalent atherosclerosis: the Dallas Heart Study. J Am Coll Cardiol. 2007 Aug 21;50(8):752-9. doi: 10.1016/j.jacc.2007.04.066. Epub 2007 Aug 6. PMID 17707180
- [Background] Cerhan JR, Moore SC, Jacobs EJ, Kitahara CM, Rosenberg PS, Adami HO, Ebbert JO, English DR, Gapstur SM, Giles GG, Horn-Ross PL, Park Y, Patel AV, Robien K, Weiderpass E, Willett WC, Wolk A, Zeleniuch-Jacquotte A, Hartge P, Bernstein L, Berrington de Gonzalez A. A pooled analysis of waist circumference and mortality in 650,000 adults. Mayo Clin Proc. 2014 Mar;89(3):335-45. doi: 10.1016/j.mayocp.2013.11.011. PMID 24582192
- [Background] Alberti KG, Zimmet P, Shaw J; IDF Epidemiology Task Force Consensus Group. The metabolic syndrome--a new worldwide definition. Lancet. 2005 Sep 24-30;366(9491):1059-62. doi: 10.1016/S0140-6736(05)67402-8. No abstract available. PMID 16182882
- [Background] Hsu WC, Araneta MR, Kanaya AM, Chiang JL, Fujimoto W. BMI cut points to identify at-risk Asian Americans for type 2 diabetes screening. Diabetes Care. 2015 Jan;38(1):150-8. doi: 10.2337/dc14-2391. No abstract available. PMID 25538311
- [Background] Neeland IJ, Ayers CR, Rohatgi AK, Turer AT, Berry JD, Das SR, Vega GL, Khera A, McGuire DK, Grundy SM, de Lemos JA. Associations of visceral and abdominal subcutaneous adipose tissue with markers of cardiac and metabolic risk in obese adults. Obesity (Silver Spring). 2013 Sep;21(9):E439-47. doi: 10.1002/oby.20135. Epub 2013 May 19. PMID 23687099
- [Background] Neeland IJ, Turer AT, Ayers CR, Powell-Wiley TM, Vega GL, Farzaneh-Far R, Grundy SM, Khera A, McGuire DK, de Lemos JA. Dysfunctional adiposity and the risk of prediabetes and type 2 diabetes in obese adults. JAMA. 2012 Sep 19;308(11):1150-9. doi: 10.1001/2012.jama.11132. PMID 22990274
- [Background] Chandra A, Neeland IJ, Berry JD, Ayers CR, Rohatgi A, Das SR, Khera A, McGuire DK, de Lemos JA, Turer AT. The relationship of body mass and fat distribution with incident hypertension: observations from the Dallas Heart Study. J Am Coll Cardiol. 2014 Sep 9;64(10):997-1002. doi: 10.1016/j.jacc.2014.05.057. PMID 25190234
- [Background] Neeland IJ, Gupta S, Ayers CR, Turer AT, Rame JE, Das SR, Berry JD, Khera A, McGuire DK, Vega GL, Grundy SM, de Lemos JA, Drazner MH. Relation of regional fat distribution to left ventricular structure and function. Circ Cardiovasc Imaging. 2013 Sep;6(5):800-7. doi: 10.1161/CIRCIMAGING.113.000532. Epub 2013 Aug 8. PMID 23929898
- [Background] Britton KA, Massaro JM, Murabito JM, Kreger BE, Hoffmann U, Fox CS. Body fat distribution, incident cardiovascular disease, cancer, and all-cause mortality. J Am Coll Cardiol. 2013 Sep 3;62(10):921-5. doi: 10.1016/j.jacc.2013.06.027. Epub 2013 Jul 10. PMID 23850922
- [Background] Wadden TA, Hollander P, Klein S, Niswender K, Woo V, Hale PM, Aronne L; NN8022-1923 Investigators. Weight maintenance and additional weight loss with liraglutide after low-calorie-diet-induced weight loss: the SCALE Maintenance randomized study. Int J Obes (Lond). 2013 Nov;37(11):1443-51. doi: 10.1038/ijo.2013.120. Epub 2013 Jul 1. PMID 23812094
- [Background] Borga M, Thomas EL, Romu T, Rosander J, Fitzpatrick J, Dahlqvist Leinhard O, Bell JD. Validation of a fast method for quantification of intra-abdominal and subcutaneous adipose tissue for large-scale human studies. NMR Biomed. 2015 Dec;28(12):1747-53. doi: 10.1002/nbm.3432. Epub 2015 Nov 2. PMID 26768490
- [Background] Schaudinn A, Linder N, Garnov N, Kerlikowsky F, Bluher M, Dietrich A, Schutz T, Karlas T, Kahn T, Busse H. Predictive accuracy of single- and multi-slice MRI for the estimation of total visceral adipose tissue in overweight to severely obese patients. NMR Biomed. 2015 May;28(5):583-90. doi: 10.1002/nbm.3286. Epub 2015 Mar 25. PMID 25808071
- [Background] Dong Z, Luo Y, Zhang Z, Cai H, Li Y, Chan T, Wu L, Li ZP, Feng ST. MR quantification of total liver fat in patients with impaired glucose tolerance and healthy subjects. PLoS One. 2014 Oct 24;9(10):e111283. doi: 10.1371/journal.pone.0111283. eCollection 2014. PMID 25343445
- [Background] Thomas MS, Newman D, Leinhard OD, Kasmai B, Greenwood R, Malcolm PN, Karlsson A, Rosander J, Borga M, Toms AP. Test-retest reliability of automated whole body and compartmental muscle volume measurements on a wide bore 3T MR system. Eur Radiol. 2014 Sep;24(9):2279-91. doi: 10.1007/s00330-014-3226-6. Epub 2014 May 29. PMID 24871333
- [Background] Human energy requirements: report of a joint FAO/ WHO/UNU Expert Consultation. Food Nutr Bull. 2005 Mar;26(1):166. No abstract available. PMID 15810802
- [Derived] Neeland IJ, Marso SP, Ayers CR, Lewis B, Oslica R, Francis W, Rodder S, Pandey A, Joshi PH. Effects of liraglutide on visceral and ectopic fat in adults with overweight and obesity at high cardiovascular risk: a randomised, double-blind, placebo-controlled, clinical trial. Lancet Diabetes Endocrinol. 2021 Sep;9(9):595-605. doi: 10.1016/S2213-8587(21)00179-0. Epub 2021 Aug 3. PMID 34358471

RESULTS

PARTICIPANT FLOW:
Groups:
- Liraglutide 3.0 mg: Drug: Liraglutide Active Drug
  Other Names:
  * Saxenda
  Escalate the liraglutide (active) dose to 3.0 mg/day over a 4 week period following an initial dose of 0.6 mg/day and weekly dose escalation steps of 0.6 mg/day through subcutaneous injection.
  Liraglutide: Liraglutide is administered once daily by subcutaneous injections with the pen-injector, either in the abdomen, thigh or upper arm. Injections can be done at any time of day irrespective of meals. Subjects will be instructed to escalate the liraglutide dose to 3.0 mg/day over a 4 week period following an initial dose of 0.6 mg/day and weekly dose escalation steps of 0.6 mg/day.
- Placebo: Drug: Placebo (for Liraglutide at a concentration of 6.0 mg/mL) Placebo tablet manufactured to mimic Liraglutide at a concentration of 6.0 mg/mL
  Other Names:
  * Placebo
  * Saline injection
  Escalate the Placebo dose to 3.0 mg/day over a 4 week period following an initial dose of 0.6 mg/day and weekly dose escalation steps of 0.6 mg/day through subcutaneous injection.
  Placebo: Placebo is administered once daily by subcutaneous injections with the pen-injector, either in the abdomen, thigh or upper arm. Injections can be done at any time of day irrespective of meals. Subjects will be instructed to escalate the placebo dose to 3.0 mg/day over a 4 week period following an initial dose of 0.6 mg/day and weekly dose escalation steps of 0.6 mg/day.
Period: Overall Study
Arm/Group | Liraglutide 3.0 mg | Placebo
Started | 92 | 93
Completed | 73 | 55
Not Completed | 19 | 38
Not completed — Lost to Follow-up | 18 | 23
Not completed — Withdrawal by Subject | 0 | 15
Not completed — Uninterpretable Outcome (Imaging) | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants analyzed if they completed an endpoint assessment and had interpretable imaging data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide 3.0 mg | Placebo | Total
Number analyzed (Participants) | 73 | 55 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (9.8) | 50.9 (8.8) | 50.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 51 | 118
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 12 | 30
  Not Hispanic or Latino | 55 | 43 | 98
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 19 | 47
  White | 43 | 35 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Total Adipose tissue [Mean (Standard Deviation); unit: Liters] | 39.6 (8.9) | 40.9 (9.8) | 40.2 (9.3)
Visceral Adipose Tissue [Mean (Standard Deviation); unit: Liters] | 4.5 (2.1) | 4.5 (1.7) | 4.5 (1.9)
Abdominal Adipose Tissue [Mean (Standard Deviation); unit: Liters] | 15.6 (4.3) | 16.2 (4.2) | 15.8 (4.2)
Lower Body Adipose Tissue [Mean (Standard Deviation); unit: Liters] — MRI based quantification of adipose tissue from the lower body.
  Liters | 14.7 (4.3) | 15.6 (5.0) | 15.1 (4.6)
Liver Fat [Mean (Standard Deviation); unit: percentage of fat] | 7.6 (7.9) | 6.1 (6.1) | 6.9 (7.2)
Total Body Lean Tissue [Mean (Standard Deviation); unit: Liters] | 21.6 (3.8) | 21.5 (3.5) | 21.5 (3.7)
Fasting Blood Glucose [Mean (Standard Deviation); unit: mg/dL] | 100.6 (12.9) | 99.1 (14.4) | 100 (13.5)
Fasting Insulin [Mean (Standard Deviation); unit: mIU/L] | 16.3 (10.8) | 18.0 (17.0) | 17.0 (13.8)
Triglycerides (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 109.4 (49.7) | 118.3 (50.6) | 113.2 (50.1)
C-reactive Protein (mg/L) [Mean (Standard Deviation); unit: mg/L] | 8.0 (4.3) | 7.8 (6.8) | 7.9 (5.6)
N-terminal prohormone of brain natriuretic peptide (NT-proBNP) (pg/mL) [Mean (Standard Deviation); unit: pg/mL] | 59.6 (44.1) | 63.2 (44.7) | 61.1 (44.1)
Number of Participants with Hypertension [Count of Participants; unit: Participants] | 30 | 20 | 50
Number of Participants with Hyperlipidemia [Count of Participants; unit: Participants] | 15 | 16 | 31
Number of Participants with Prediabetes [Count of Participants; unit: Participants] | 2 | 3 | 5
Systolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 130.3 (14.9) | 125.8 (13.9) | 128.4 (14.6)
Diastolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 80.9 (7.8) | 78.5 (8.3) | 79.8 (8.1)
Weight (kg) [Mean (Standard Deviation); unit: Kg] | 101.0 (17.9) | 102.3 (17.9) | 101.5 (17.9)
Height (m) [Mean (Standard Deviation); unit: m] | 1.6 (0.1) | 1.6 (0.1) | 1.6 (0.1)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 37.2 (6.0) | 38.1 (6.1) | 37.6 (6.1)
Waist Circumference (cm) [Mean (Standard Deviation); unit: cm] | 105.5 (12.2) | 104.8 (10.6) | 105.2 (11.5)
Baseline kcal/day [Mean (Standard Deviation); unit: kcal/day] | 2177 (195) | 2196 (189) | 2185 (192)

OUTCOME MEASURES:

1. Primary Outcome: Relative Percent Reduction in Visceral Adipose Tissue Mass Measured by MRI
Description: The effect on relative percent reduction from baseline in visceral adipose tissue mass measured by MRI after 40 weeks on treatment.
  Positive numbers reflect the reduction in the value from baseline to study endpoint as a percent of the baseline.
  Reduction in this variable is believed to be associated with lower cardiovascular risk.
Time Frame: Baseline, 40 weeks
Population: Those who completed study endpoint assessment (interpretable MRI at baseline and at study end).
Measure: Mean (95% Confidence Interval); unit: percentage of reduction in VAT
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
percentage of reduction in VAT | 12.49 [10.4 to 14.6] | 1.63 [-1.62 to 4.88]

2. Secondary Outcome: Absolute Reduction in Visceral Adipose Tissue Volume
Description: The effect on absolute reduction from baseline in visceral adipose tissue mass measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
  Reduction in this variable is believed to be associated with lower cardiovascular risk.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
Liters | 0.53 (0.43) | 0.10 (0.53)

3. Secondary Outcome: Relative Percent Reduction in Body Weight
Description: The effect on relative percent reduction from baseline in body weight after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
  Reduction in this variable is believed to be associated with lower cardiovascular risk.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
percent change | 6.59 (4.80) | 1.19 (4.68)

4. Secondary Outcome: Absolute Reduction in Body Weight
Description: The effect on absolute reduction from baseline in body weight after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
  Reduction in this variable is believed to be associated with lower cardiovascular risk.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
Kilograms | 6.75 (5.35) | 1.3 (4.79)

5. Secondary Outcome: Relative Percent Reduction in Waist Circumference
Description: The effect on relative percent reduction from baseline in waist circumference after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
  Reduction in this variable is believed to be associated with lower cardiovascular risk.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
percent change | 6.90 (6.43) | 4.16 (6.06)

6. Secondary Outcome: Absolute Reduction in Waist Circumference
Description: The effect on absolute reduction from baseline in waist circumference after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
  Reduction in this variable is believed to be associated with lower cardiovascular risk.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
cm | 7.4 (6.8) | 4.6 (6.7)

7. Secondary Outcome: Relative Percent Reduction in Total Body Adipose Tissue
Description: The effect on relative percent reduction from baseline in total body adipose tissue (fat) mass measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
  Reduction in this variable is believed to be associated with lower cardiovascular risk.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
percent change | 9.59 (7.15) | 0.95 (7.80)

8. Secondary Outcome: Absolute Reduction in Total Body Adipose Tissue
Description: The effect on absolute reduction from baseline in total body adipose tissue mass measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
  Reduction in this variable is believed to be associated with lower cardiovascular risk.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
Liters | 3.76 (2.87) | 0.42 (2.92)

9. Secondary Outcome: Relative Percent Reduction in Abdominal Subcutaneous Adipose Tissue
Description: The effect on relative percent reduction from baseline in abdominal subcutaneous adipose tissue mass measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
percent change | 9.87 (8.23) | 0.77 (8.40)

10. Secondary Outcome: Absolute Reduction in Abdominal Subcutaneous Adipose Tissue
Description: The effect on absolute reduction from baseline in abdominal subcutaneous adipose tissue mass measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
Liters | 1.52 (1.31) | 0.15 (1.24)

11. Secondary Outcome: Relative Percent Reduction in Lower Body Subcutaneous Adipose Tissue
Description: The effect on relative percent reduction from baseline in lower body subcutaneous adipose tissue mass measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
percent change | 9.95 (7.61) | 1.29 (8.57)

12. Secondary Outcome: Absolute Reduction in Lower Body Subcutaneous Adipose Tissue
Description: The effect on absolute reduction from baseline in lower body subcutaneous adipose tissue mass measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
Liters | 1.51 (1.34) | 0.19 (1.19)

13. Secondary Outcome: Relative Percent Reduction in Liver Fat Percent
Description: The effect on relative percent reduction from baseline in liver (hepatic) fat percentage measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint. Negative values reflect an increase in the value from baseline to study endpoint.
  Reduction in this variable is believed to be associated with lower cardiovascular risk.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
percent change | 12.37 (61.43) | -20.63 (104.92)

14. Secondary Outcome: Absolute Reduction in Liver Fat Percent
Description: The effect on absolute reduction from baseline in liver (hepatic) fat percentage measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint. Negative values reflect an increase in the value from baseline to study endpoint.
  Reduction in this variable is believed to be associated with lower cardiovascular risk.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images are reported here.
Measure: Mean (Standard Deviation); unit: percentage of liver fat
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
percentage of liver fat | 2.35 (5.35) | -0.01 (3.24)

15. Secondary Outcome: Relative Percent Reduction in Total Body Lean Volume
Description: The effect on relative percent reduction from baseline in total body lean volume (fat-free mass) measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images are reported here.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
percent change | 2.47 (4.04) | 0.90 (3.66)

16. Secondary Outcome: Absolute Reduction in Total Body Lean Volume
Description: The effect on absolute reduction from baseline in total body lean volume (fat-free mass) measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images are reported here.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
Liters | 0.54 (0.88) | 0.17 (0.80)

17. Secondary Outcome: Relative Percent Reduction in Total Thigh Muscle Volume
Description: The effect on relative percent reduction from baseline in total thigh muscle volume measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images are reported here.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
percent change | 3.48 (3.55) | 0.68 (3.72)

18. Secondary Outcome: Absolute Reduction in Total Thigh Muscle Volume
Description: The effect on absolute reduction from baseline in total thigh muscle volume measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
Time Frame: Baseline, 40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images are reported here.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
Liters | 0.35 (0.35) | 0.06 (0.38)

19. Secondary Outcome: Relative Percent Reduction in Mean Anterior Thigh Muscle Fat Infiltration Percent
Description: The effect on relative percent reduction from baseline in mean anterior thigh muscle fat infiltration percent measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint. Negative values reflect an increase in the value from baseline to study endpoint.
  Reduction in this variable is believed to be associated with lower risk for metabolic disease.
Time Frame: Baseline,40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images are reported here.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
percent change | 2.81 (6.51) | -0.29 (6.96)

20. Secondary Outcome: Absolute Reduction in Mean Anterior Thigh Muscle Fat Infiltration Percent
Description: The effect on absolute reduction from baseline in mean anterior thigh muscle fat infiltration percent measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint. Negative values reflect an increase in the value from baseline to study endpoint.
  Reduction in this variable is believed to be associated with lower risk for metabolic disease
Time Frame: Baseline,40 weeks
Population: Those who completed baseline and endpoint MRI with interpretable images are reported here.
Measure: Mean (Standard Deviation); unit: percentage of fat infiltration
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
percentage of fat infiltration | 0.23 (0.49) | 0.01 (0.58)

21. Secondary Outcome: Change From Baseline in VAT/SAT Ratio
Description: The effect on absolute reduction from baseline in Visceral adipose tissue/subcutaneous adipose tissue (VAT/SAT) ratio measured by MRI after 40 weeks on treatment versus placebo.
  Positive numbers reflect the reduction in the value from baseline to study endpoint.
  This is the ratio of visceral adipose tissue to subcutaneous adipose tissue and it is thought that lower values (relatively less visceral adipose tissue) are better.
Time Frame: Baseline, 40 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
ratio | 0.01 (0.03) | 0 (0.02)

22. Secondary Outcome: Change From Baseline in Total Fat/Fat-free Mass Ratio
Description: The effect on absolute change from baseline in total fat/fat-free mass ratio measured by MRI after 40 weeks on treatment versus placebo.
  This is a ratio of fat to lean mass and it is believed that lower values (less fat relative to lean mass) is better.
Time Frame: Baseline, 40 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
ratio | -7.23 (7.25) | 0.01 (7.83)

23. Secondary Outcome: Relative Percent Change in Fasting Blood Glucose
Description: The relative percent change in fasting blood glucose from baseline to study end point as a percent of baseline by treatment group.
  Negative values reflect a reduction. This is a blood based biomarker for diabetes in which normal levels are desirable (70-100 mg/dL).
Time Frame: Baseline, 40 weeks
Population: Complete case analysis was done. Those who completed baseline and endpoint study visits and had results, were only analyzed and reported here.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
percent change | -5.62 (10.77) | 0.83 (13.31)

24. Secondary Outcome: Relative Percent Change in Insulin
Description: The relative percent change in insulin from baseline to study end point as a percent of baseline by treatment group.
  Positive values reflect an increase. Collection was impacted by coronavirus disease 2019 (COVID-19) and limitations to in person study visits, limiting complete collection of data for this measure.
  This is a blood based biomarker in which lower fasting levels are desirable.
Time Frame: Baseline, 40 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 72 | 54
percent change | 20.58 (70.69) | 7.73 (58.09)

25. Secondary Outcome: Relative Percent Change in HOMA-IR
Description: The relative percent change in HOMA-IR from baseline to study end point as a percent of baseline by treatment group.
  Positive values reflect an increase. Collection was impacted by coronavirus disease 2019 (COVID-19) and limitations to in person study visits, limiting complete collection of data for this measure.
  The relative percent change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) from baseline to study end point by treatment group measures insulin resistance. Levels above 1.9 signal early insulin resistance, while levels above 2.9 signal significant insulin resistance. There will be optimal insulin sensitivity if HOMA-IR is less than 1.
Time Frame: Baseline, 40 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 72 | 54
percent change | 15.35 (71.44) | 11.85 (69.0)

26. Secondary Outcome: Relative Percent Change in C-reactive Protein
Description: The relative percent change in biomarker of inflammation: C-reactive protein (CRP) from baseline to study end point as a percent of baseline by treatment group.
  Negative values reflect a decrease. Collection was impacted by coronavirus disease 2019 (COVID-19) and limitations to in person study visits, limiting complete collection of data for this measure.
  This is a blood based test for which lower values are associated with less inflammation and lower risk for cardiovascular events.
Time Frame: Baseline, 40 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 27 | 30
percent change | -19.91 (32.75) | 19.02 (76.13)

27. Secondary Outcome: Relative Percent Change in Triglyceride/HDL-C Ratio
Description: The relative percent change in triglyceride/HDL-C ratio from baseline to study end point as a percent of baseline by treatment group.
  Negative values reflect a decrease. Collection was impacted by coronavirus disease 2019 (COVID-19) and limitations to in person study visits, limiting complete collection of data for this measure.
  Lower ratio of triglycerides to HDL-cholesterol is associated with less insulin resistance and lower cardiovascular risk.
Time Frame: Baseline, 40 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 42 | 32
percent change | -2.10 (30.23) | -2.18 (28.97)

28. Secondary Outcome: Relative Percent Change in Nt-proBNP
Description: The relative percent change in N-terminal Pro Brain Natriuretic Peptides (Nt-proBNP) from baseline to study end point as a percent of baseline by treatment group.
  Negative values reflect a decrease. Collection was impacted by coronavirus disease 2019 (COVID-19) and limitations to in person study visits, limiting complete collection of data for this measure.
  NT-proBNP is a blood based biomarker. Lower levels are associated with lower risk for heart failure and cardiovascular events.
Time Frame: Baseline, 40 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 58 | 40
percent change | 12.10 (78.5) | 20.47 (79.42)

29. Secondary Outcome: Absolute Change in Fasting Blood Glucose
Description: The change in fasting blood glucose from baseline to study end point by treatment group.
Time Frame: Baseline,40 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
mg/dL | -6.49 (12.41) | -0.22 (12.93)

30. Secondary Outcome: Absolute Change in Insulin
Description: The absolute change in insulin from baseline to study end point by treatment group. Collection was impacted by COVID-19 and changes to study visits.
Time Frame: Baseline, 40 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 72 | 54
mIU/L | 0.75 (9.67) | -1.48 (12.26)

31. Secondary Outcome: Absolute Change in HOMA-IR
Description: The absolute change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) from baseline to study end point by treatment group measures insulin resistance. Levels above 1.9 signal early insulin resistance, while levels above 2.9 signal significant insulin resistance. There will be optimal insulin sensitivity if HOMA-IR is less than 1. Collection was impacted by COVID-19 and changes to study visits.
Time Frame: Baseline, 40 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Molar units
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 72 | 54
Molar units | -0.15 (3.15) | -0.69 (5.24)

32. Secondary Outcome: Absolute Change in CRP
Description: The change in Markers of inflammation: C-reactive protein (CRP) from baseline to study end point by treatment group. Collection was impacted by COVID-19 and changes to study visits.
  This is a blood based test for which lower values are associated with less inflammation and lower risk for cardiovascular events.
Time Frame: Baseline, 40 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 27 | 30
mg/L | -2.18 (3.37) | -0.64 (6.23)

33. Secondary Outcome: Absolute Change in Triglyceride/HDL-C Ratio
Description: The change in triglyceride/HDL-C ratio from baseline to study end point by treatment group. Collection was impacted by COVID-19 and changes to study visits.
  Lower ratio of triglycerides to HDL-cholesterol is associated with less insulin resistance and lower cardiovascular risk.
Time Frame: Baseline, 40 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 42 | 32
ratio | -0.02 (0.83) | -0.16 (0.69)

34. Secondary Outcome: Absolute Change in Nt-proBNP
Description: The change in N-terminal Pro Brain Natriuretic Peptides (Nt-proBNP) from baseline to study end point by treatment group. Collection was impacted by COVID-19 and changes to study visits.
  NT-proBNP is a blood based biomarker. Lower levels are associated with lower risk for heart failure and cardiovascular events.
Time Frame: Baseline, 40 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 58 | 40
pg/mL | -8.10 (48.82) | 1.44 (41.04)

35. Secondary Outcome: Change From Baseline in Heart Rate
Description: The change in heart rate/pulse from baseline to study endpoint visit by treatment group.
Time Frame: Baseline, 40 weeks
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
beats per minute | 4.84 (12.95) | 2.67 (11.39)

36. Secondary Outcome: Change From Baseline in Blood Pressure
Description: The change in systolic blood pressure from baseline to study endpoint visit by treatment group.
Time Frame: Baseline, 40 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
mmHg | -5.84 (17.98) | -0.02 (16.01)

37. Other Pre Specified Outcome: On-treatment Time, Weeks
Description: The mean duration of treatment during study follow-up.
Time Frame: weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 55
weeks | 36.2 (8.6) | 36.1 (8.2)

ADVERSE EVENTS:
Time Frame: For the entire duration of the study: 40 weeks.
Description: Adverse events collected at each study visit. GI side effects captured and reported in summary form.
Arm/Group | Liraglutide 3.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/93
Other Adverse Events (participants affected / at risk) | 53/92 | 34/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 3.0 mg (N=92) | Placebo (N=93)
GI related (Gastrointestinal disorders) | 43 (43) | 12 (12) — Constipation, nausea/vomiting, upset stomach, diarrhea
Respiratory Tract infection (Infections and infestations) | 10 (10) | 14 (14) — Upper Respiratory Infection (URI) or pharyngitis
Injection site reaction (Product Issues) | 7 (7) | 8 (8)
headache (Nervous system disorders) | 5 (5) | 5 (5)
joint pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
insomnia (Nervous system disorders) | 2 (2) | 0 (0)
dizziness (Nervous system disorders) | 3 (3) | 0 (0)
fever (Immune system disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Results reported according to updated statistical analysis plan published 7/28/2020 on CT.gov website. The updated 7/28/2020 analysis plan accounted for changes in data collection (blood biomarkers) during COVID-19 pandemic and was submitted and published prior to study completion and prior to study un-blinding with updated terminology for study endpoints compared to original protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT03038620/Prot_001.pdf
  • Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT03038620/SAP_002.pdf